CLINICAL TRIAL: NCT06363227
Title: Postoperative Pain After Implementation of Standardized Pain Therapy Management in Orthopaedic Patients A Quality Assessment in Major Orthopaedic and Spine Surgery
Brief Title: Postoperative Pain After Implementation of Standardized Pain Therapy Management in Orthopaedic Patients
Acronym: PAIN
Status: Not yet recruiting | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Christoph Hofer, Head of Anesthesia, Professor, Principal Investigator, Schulthess Klinik
Other Study IDs: ANEST-0003
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain, Acute
Keywords: multimodal pain protocol; orthopedic surgery; opioids
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Standardized pain management — multimodal postoperative pain protocol

SUMMARY:
The aim of this study is to examine the impact of implementing a standardized pain therapy protocol and their components on postoperative pain trajectories and postoperative outcomes such as increased opioid consumption and to compare it for different orthopaedic operations, i.e. major shoulder, hip, knee und spine surgery.

DETAILED DESCRIPTION:
A multimodal standardized pain management was implemented at the Schulthess Clinic in 2002, followed by the gradual introduction of a standardized ultrasound-guided perioperative regional anaesthesia program. Along with these measures, an improved preoperative screening process for patients at risk of increased post-operative pain has been installed and an improved individual pain assessment in the perioperative period has been introduced. This allowed for the creation of pain trajectories, which the pain team started to use to identify gaps in the management of different patient groups. An example of a trajectory group is shown in Figure 1. These pain trajectories have not yet been evaluated for the overall implementation cycle of the multimodal standardized pain management in order to further improve postoperative care especially for patients with a history of chronic pain and those prone to opioid overconsumption.We hypothesise that pain trajectories have changed significantly over the study period as standardised pain management has been implemented. We also hypothesise that patients with chronic pain and increased opioid consumption will have different pain trajectories compared to all other patients. However, we believe that the pain trajectories for different orthopaedic surgeries do not show much variation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary hip and knee arthroplasties or revision surgery:CHOP Code: 81.51, 81.52, 81.52, 81.54
* Patients undergoing primary shoulder or revision surgery: CHOP codes: 81.80.11, 81.80.12, 83.64.11, 81.82.35, 81.82.45, 81.82.46, 81.82.47
* Patients undergoing major spine surgery: CHOP Code: 7A.6, 7A.7

Exclusion Criteria:

- Patients who did not sign general informed consent (for the Schulthess Clinic).

Ages: 16 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective major orthopedic or spine surgery at the Schulthess Clinic between 2020 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Perioperative pain trajectories | 2021-2024
  Pain scores based on perioperative NRS = Numeric rating scales (0-10) prior to surgery on day of admission and during the postoperative period until discharge
Increased risk for postoperative pain | 2021-2024
  Identification of risk factors

SECONDARY OUTCOMES:
Total amount of opioids administered | 2021-2024
  iv and po opioids given in the postoperative period
Correlation of pain trajectories and patient reported outcome measures (e.g. postoperative nausea and vomiting) | 2021-2024

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Hofer, MD, Principal Investigator — Schulthess Klinik